CLINICAL TRIAL: NCT03775616
Title: Development of a Comprehensive Financial Navigation Program for Patients With Cancer and Their Caregivers
Brief Title: Financial Navigation Program Intervention in Supporting Patients With Solid Tumors and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1001593; NCI-2018-02607 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 8570 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-12-10; First posted 2018-12-14 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Caregiver; Solid Neoplasm
MeSH Terms: interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive (financial navigation program) (Experimental): Participants receive financial navigation program intervention consisting of a financial navigation video, monthly one-one financial counselling session, monthly phone or email consultation with patient navigators for 6 months and complete surveys at baseline, 3, 6, and 12 months.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Educational Intervention — Receive financial navigation program intervention
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This trial studies how well a financial navigation program intervention works in supporting patients with solid tumors and their caregivers. The financial navigation program intervention is an educational course about cancer treatment cost. This educational course may provide cancer patients and their caregivers with helpful information about dealing with cancer treatment cost.

DETAILED DESCRIPTION:
Participants receive financial navigation program intervention consisting of a financial navigation video, monthly one-one financial counselling session, monthly phone or email consultation with patient navigators for 6 months and complete surveys at baseline, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: Any solid tumor diagnosis (any stage)
* PATIENTS: Currently receiving (or completed within 6 months) chemotherapy, radiation, or hormonal therapy for cancer
* PATIENTS: In the treating physician's best estimation, has a life expectancy of 6 months or greater
* PATIENTS: Able to identify a primary caregiver who is involved in helping with the logistics, financial, or emotional aspects of his/her cancer care
* PATIENTS: English-speaking
* CAREGIVERS: Caregiver of a patient who is eligible for to participate in the study
* CAREGIVERS: English-speaking

Exclusion Criteria:

* PATIENTS: Cognitive or other impairment that would interfere with ability to understand and/or respond to questions about personal finances and paying for cancer treatment
* PATIENTS: Hematologic malignancy (e.g. multiple myeloma, lymphoma, leukemia)
* CAREGIVERS: cognitive or other impairment that would interfere with ability to understand and/or respond to questions about patient fiances and paying for cancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Accrual rate (number of patients and caregivers enrolled per month) | Up to 12 months
Time to accrual | Up to 12 months
Proportion of participants completing each of the 3 program components | Up to 12 months
Proportion of participants completing the entire program and 6 month follow up | Up to 6 months
Financial status assessment | Up to 12 months
  Prior to and following participation in the financial navigation program, patients will complete questionnaire and provide basic information about their financial status including household income, assets, educational level, and employment status.
Financial distress assessment questionnaire | Up to 12 months
  Will measure patients' level of financial distress before and after participation in various components of the program via a questionnaire that indicates financial distress based on responses
Patient advocate foundation (PAF) navigators | Up to 12 months
  PAF navigators will tract all issues identified during an initial need assessment with the patients and subsequently all outcomes of any such issues.
Consumer education and training services (CENTS) financial counselors | Up to 12 months
  The CENTs financial counselors will tract specific recommendations given each patient during the course of the study and share these recommendation with the investigators.
Family Reach staff feedback | Up to 12 months
  Family Reach will track patients that have been granted financial assistance, and will provide any further information obtained from patients interaction.

CONTACTS AND LOCATIONS:
Overall Officials: Veena Shankaran, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No